CLINICAL TRIAL: NCT05107219
Title: Pilot Study of GCC Agonists to Identify a Cyclic-GMP Signal in Duodenal Tissue of Volunteers
Brief Title: GCC Agonist Signal in the Small Intestine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2021-11620; NCI-2021-11620 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UWI21-06-01 (Other: University of Wisconsin Carbone Cancer Center - University Hospital); UWI21-06-01 (Other: DCP); P30CA014520 (NIH); UG1CA242635 (NIH)
Record Dates: First submitted 2021-11-03; First posted 2021-11-04 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-05

CONDITIONS: Barrett Esophagus; Gastroesophageal Reflux Disease; Malignant Digestive System Neoplasm
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Gastrointestinal Neoplasms | interventions — Biopsy; Specimen Handling; Endoscopy, Digestive System; linaclotide; plecanatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (plecanatide, EGD) (Experimental): Patients receive a single dose of plecanatide (3 mg) PO 60-120 minutes prior to standard of care EGD with biopsy and luminal fluid collection.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Esophagogastroduodenoscopy; Drug: Plecanatide
- Arm II (linaclotide, EGD) (Experimental): Patients receive a single dose of linaclotide (145 mcg) PO 60-120 minutes prior to standard of care EGD with biopsy and luminal fluid collection.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Esophagogastroduodenoscopy; Drug: Linaclotide
- Arm III (EGD) (Active Comparator): Patients undergo standard of care EGD with biopsy and luminal fluid collection.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Esophagogastroduodenoscopy

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of luminal fluid
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Esophagogastroduodenoscopy — Undergo EGD
  Other Names: EGD
Drug: Linaclotide — Given PO
  Other Names: [9-L-tyrosine]heat-stable enterotoxin (Escherichia coli)-(6-19)-peptide; Linzess; MD-1100
  Arms: Arm II (linaclotide, EGD)
Drug: Plecanatide — Given PO
  Other Names: Trulance
  Arms: Arm I (plecanatide, EGD)

SUMMARY:
This early phase I trial studies the guanylyl cyclase C (GCC) agonist effect on cGMP signal in duodenal tissue. Plecanatide and linaclotide are drugs approved by the Food and Drug Administration for the treatment of conditions related to constipation. This trial aims to see the effects of taking either one of two drugs, plecanatide or linaclotide, or no drug, on a certain chemical found in the tissue collected from small intestine and how they compare.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess and compare participants randomly assigned 1:1:1 to one of three intervention arms (plecanatide 3 mg versus linaclotide 145 mcg versus no active agent) with respect to change in cyclic guanosine monophosphate (cGMP) accumulation in normal appearing duodenal mucosa specimens.

SECONDARY OBJECTIVES:

I. Characterization and comparison of the following outcomes (in prioritized order):

Ia. cGMP levels in luminal fluid from participants receiving either linaclotide or plecanatide to fluid from participants receiving no agent; Ib. Vasodilator stimulated phosphoprotein (VASP) phosphorylation in normal-appearing duodenal mucosa biopsy specimens from participants receiving either linaclotide or plecanatide to those specimens from participants receiving no agent.

EXPLORATORY OBJECTIVES:

I. Comparison of cGMP and VASP phosphorylation between the plecanatide and linaclotide arms.

II. Transcriptome analysis of cellular response (ribonucleic acid [RNA] sequencing analyses) to define whether GCC ligand exposure induces reproducible changes in duodenal messenger [m]RNA expression that can serve as a reliable biomarker of GCC-cGMP signaling in future studies.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive a single dose of plecanatide (3 mg) orally (PO) 60-120 minutes prior to standard of care esophagogastroduodenoscopy (EGD) with biopsy and luminal fluid collection. Patients also undergo biopsy on study.

ARM II: Patients receive a single dose of linaclotide (145 mcg) PO 60-120 minutes prior to standard of care EGD with biopsy and luminal fluid collection. Patients also undergo biopsy on study.

ARM III: Patients undergo standard of care EGD with biopsy and luminal fluid collection. Patients also undergo biopsy on study.

After completion of study intervention, patients are followed up at day 7.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for clinically indicated esophagogastroduodenoscopy (EGD)
* Age >= 18 years of age. Note: Because no dosing or adverse event (AE) data are currently available on the use of plecanatide or linaclotide in participants < 18 years of age, children and adolescents are excluded from this study but will be eligible for future pediatric trials, if applicable
* Willing to provide mandatory biospecimens as specified in the protocol
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Not pregnant or breastfeeding, as determined by pregnancy test prior to EGD procedure. Note: The effects of plecanatide and linaclotide on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 2 weeks after discontinuing study agent. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately. Breastfeeding should be discontinued if the mother is treated with plecanatide or linaclotide
* Ability to understand and the willingness to sign a written informed consent document
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients on chronic suppressive antiviral therapy for herpes simplex virus (HSV) are eligible

Exclusion Criteria:

* Prior treatment in the past week with plecanatide, linaclotide, or other agent whose primary mechanism of action is that of a GCC agonist
* History of allergic reactions attributed to compounds of similar chemical or biologic composition of plecanatide or linaclotide
* Use of any other investigational agents =< 12 weeks prior to registration
* Uncontrolled intercurrent illness, or psychiatric illness/social situations that would limit compliance with study requirements
* History of gastric bypass, gastric sleeve, or bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Cyclic guanosine monophosphate (cGMP) levels | Up to 2 years
  Will compare cGMP levels measured in normal-appearing duodenal mucosa biopsy specimens from participants receiving linaclotide or plecanatide to cGMP levels in specimens from participants receiving no active treatment. Will evaluate the difference between the control and each treated arm in cGMP levels using two-tailed two-sample Student t-tests. If necessary, a log transformation or Wilcoxon rank-sum will be used, as appropriate.

SECONDARY OUTCOMES:
cGMP levels in luminal fluid | Up to 2 years
Vasodilator-stimulated phosphoprotein (VASP) phosphorylation in normal appearing duodenal mucosa | Up to 2 years

OTHER OUTCOMES:
Comparison pf cGMP and VASP phosphorylation between the plecanatide and linaclotide arms | Up to 2 years
Cellular response | Up to 2 years
  Transcriptome analysis of cellular response (ribonucleic acid [RNA] sequencing analyses), to define whether guanylyl cyclase C (GCC) ligand exposure induces reproducible changes in duodenal messenger (m)RNA expression that can serve as a reliable biomarker of GCC-cGMP signaling in future studies.

CONTACTS AND LOCATIONS:
Overall Officials: David S Weinberg, Principal Investigator — Fox Chase Cancer Center
Locations (4):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm